CLINICAL TRIAL: NCT00983658
Title: A Phase II, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy, Safety, and Tolerability of Intravenous huMAb OX40L (RO4989991) in the Prevention of Allergen-Induced Airway Obstruction in Adults With Mild Allergic Asthma
Brief Title: A Study of huMAb OX40L in the Prevention of Allergen-Induced Airway Obstruction in Adults With Mild Allergic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OXF4696g
Record Dates: First submitted 2009-09-21; First posted 2009-09-24 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Asthma
Keywords: Anti-OX40L; Mild Allergic Asthma; Allergies; Allergic Asthma; Adult Asthma
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- huMAb OX40L (Experimental)
  Interventions: Drug: huMAb OX40L
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: huMAb OX40L — Intravenous repeating dose
  Arms: huMAb OX40L
Drug: placebo — Intravenous repeating dose
  Arms: Placebo

SUMMARY:
This Phase II, double-blind, placebo-controlled, randomized, parallel-group study is designed to evaluate the efficacy, safety, and tolerability of huMAb OX40L administered to patients by IV infusion for the treatment of allergen-induced asthma.

ELIGIBILITY:
Inclusion Criteria:

* Weight between 50 and 125 kg
* Mild, stable allergic asthma
* History of episodic wheeze and shortness of breath
* FEV1 at baseline ≥ 70% of the predicted value
* For women of childbearing potential, agreement to use an effective means of contraception while enrolled in the study
* For men with partners of childbearing potential, willingness to use condoms with spermicide during treatment
* Ability to comprehend and follow all required study procedures
* Positive skin prick test to common aeroallergens (e.g., cat, dust, mite, grass, and pollen)
* Positive allergen-induced early and late airway bronchoconstriction

Exclusion Criteria:

* A worsening of asthma or a respiratory tract infection within 6 weeks preceding study entry
* Acute infection (including viral infection) within the 6 weeks preceding dosing (8 weeks for respiratory infections) or any ongoing chronic infection
* History of recurrent bacterial infection as an adult or history or presence of any chronic infectious condition, including (but not limited to), tuberculosis, parasitic infection, etc.
* Lung disease other than mild allergic asthma
* History of heart, lung, kidney, liver, neurologic or chronic infectious disease
* Concomitant disease or condition, which could interfere with the conduct of the study, including, but not limited to, cancer, alcoholism, drug dependency or abuse, or psychiatric disease
* History of serious adverse reaction or hypersensitivity to any drug
* Pregnancy or lactation or positive serum pregnancy test at screening
* Chronic use of any other medication for treatment of allergic lung disease other than short-acting β2-agonists or ipratropium bromide
* Current (or history of) treatment with a monoclonal antibody or chimeric biomolecule within the past 5 months (5 half-lives of the drug), including omalizumab
* Regular use of tobacco products of any kind or within the previous 6 months, or smoking history > 10 pack-years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the late asthmatic response (LAR) in patients treated with huMAb OX40L versus placebo | 16 weeks after the first dose

SECONDARY OUTCOMES:
LAR after the allergen challenge in patients treated with huMAb OX40L versus placebo | Approximately Day 56 prior to third dose
Change in methacholine challenge response relative to the pre-allergen challenge PC20 | 24 hours after each allergen challenge
Early asthmatic response (EAR) in patients treated with huMAb OX40L versus placebo | Between 0 and 2 hours after each allergen challenge
Incidence and nature of treatment-emergent adverse events | Through study completion or early study discontinuation
Incidence and nature of infusion reactions | Through study completion or early study discontinuation
Incidence of infectious complications | Through study completion or early study discontinuation
Incidence, nature, relatedness, and severity of adverse events | Through study completion or early study discontinuation
Clinically significant changes in vital signs, electrocardiograms, FEV1, and safety laboratory measures | Through study completion or early study discontinuation
Incidence of anti-therapeutic antibodies | Through study completion or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Dana McClintock, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Gauvreau GM, Boulet LP, Cockcroft DW, FitzGerald JM, Mayers I, Carlsten C, Laviolette M, Killian KJ, Davis BE, Larche M, Kipling C, Dua B, Mosesova S, Putnam W, Zheng Y, Scheerens H, McClintock D, Matthews JG, O'Byrne PM. OX40L blockade and allergen-induced airway responses in subjects with mild asthma. Clin Exp Allergy. 2014 Jan;44(1):29-37. doi: 10.1111/cea.12235. PMID 24224471